CLINICAL TRIAL: NCT03146338
Title: Prophylaxis of Magnesium-rich Mineral Water to Prevent Hypomagnesemia Induced by an Anti-EGFR Monoclonal Antibody
Brief Title: Prophylaxis of Magnesium-rich Mineral Water to Prevent Hypomagnesemia Induced by an Anti-EGFR (OPTIMAG)
Acronym: OPTIMAG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Weprom (Other)
Collaborators: Neptune (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ILC-2-2016; 2016-A01091-50 (Other: French Health Products Safety Agency)
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Metastatic Colorectal Cancer; Metastatic Head and Neck Cancer
Keywords: Anti-EGFR; Hypomagnesemia; Magnesium-rich mineral water; Metastatic colorectal or head and neck cancers
MeSH Terms: conditions — Colorectal Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium-rich mineral water (Rozana) (Experimental): Patients in this arm must take 1.5 Liter by day of a mineral water rich in magnesium (Rozana) during the treatment by anti-EGFR. The mineral water is provided.
  Interventions: Other: Magnesium-rich mineral water (Rozana)
- Standard (No Intervention): Patients will have the usual care (oral advice only according to the habits of the investigator)

INTERVENTIONS:
Other: Magnesium-rich mineral water (Rozana) — intakes of 1.5 L by day
  Arms: Magnesium-rich mineral water (Rozana)

SUMMARY:
Anti-EGFR (Epidermal Growth Factor Receptor) therapies, namely cetuximab and panitumumab, have become standards in the management of metastatic colorectal and head and neck cancers. These therapies are used in daily practice, that requiring to manage their skin and digestive toxicities. However, anti-EGFR are also frequently responsible for hypomagnesemia often neglected and under-treated.

Hypomagnesemia may manifest as asthenia, cramps, muscle weakness, mood disorders. She is often underestimated because they are difficult to identify and accountable by clinicians in the context of cancer under chemotherapy.

There is currently no national or international recommendation on the management of hypomagnesaemia in oncology and medicine in general. There are, however, on the market many nutritional supplements rich in magnesium in the form of tablets or oral solution, in multiple dosages.

These food supplements rich in magnesium are sold without proof of effectiveness. Moreover, the prescription of oral magnesium supplementation adds to the oncology patient an over-medicalization, which can be poorly tolerated at the digestive level, and responsible for diarrhea and a lack of compliance.

The European Food Safety Authority (EFSA) recommends in its opinion on "Dietary reference values for water" to consume 2 liters for women and 2.5 liters for men every day, all sources combined (food and beverages). The drink represent 80% of the water intake, that is about 1.5 Liter per day excluding food. However, there are multiple water marketed or distributed freely, with different compositions. Thus the quantity and quality of the mineral water consumed can influence the metabolism. Rozana® mineral water, has the double advantage of being the French water the most concentrated in magnesium (160 mg / L) and of being lowly concentrated in sulphate, responsible of the laxative power of certain waters.

Instead of adding magnesium supplements with a poor digestive tolerance, to patients with metastatic cancer and often with a heavy treatment , the aim of this study is to evaluate whether a change in oral hydration in quantitative and qualitative terms can decrease the rate of hypomagnesemia in patients treated with anti-EGFR.

DETAILED DESCRIPTION:
Anti-EGFR (Epidermal Growth Factor Receptor) therapies, namely cetuximab and panitumumab, have become standards in the management of metastatic colorectal and head and neck cancers. These therapies are used in daily practice, that requiring to manage their skin and digestive toxicities. However, anti-EGFR are also frequently responsible for hypomagnesemia often neglected and under-treated.

Magnesium remains the fourth cation and the second most important intracellular cation in the body. It is an indispensable cofactor in multiple enzymatic reactions. Hypomagnesemia may manifest as asthenia, cramps, muscle weakness, mood disorders. She is often underestimated because they are difficult to identify and accountable by clinicians in the context of cancer under chemotherapy.

There is currently no national or international recommendation on the management of hypomagnesaemia in oncology and medicine in general. Hypomagnesemia is, in daily practice, mostly undiagnosed or untreated. There are, however, on the market many nutritional supplements rich in magnesium in the form of tablets or oral solution, in multiple dosages.

To date, these food supplements rich in magnesium are sold without proof of effectiveness. The clinical data are very insufficient, and no oral supplementation is reimbursed. Moreover, the prescription of oral magnesium supplementation, often several intakes a day, adds to the oncology patient an over-medicalization, which can be poorly tolerated at the digestive level, and responsible for diarrhea and a lack of compliance. Oral hydration is one of the most prescribed medical advice and remains essential to combat the risk of dehydration in extreme ages. The European Food Safety Authority (EFSA) recommends in its opinion on "Dietary reference values for water" to consume 2 liters for women and 2.5 liters for men every day, all sources combined (food and beverages). The drink represent 80% of the water intake, that is about 1.5 Liter per day excluding food. However, there are multiple water marketed or distributed freely, with different compositions. Thus the quantity and quality of the mineral water consumed can influence the metabolism.

The digestive absorption of magnesium provided by mineral water in a healthy individual was evaluated at around 40 to 50%. Rozana® mineral water, has the double advantage of being the French water the most concentrated in magnesium (160 mg / L) and of being lowly concentrated in sulphate, responsible of the laxative power of certain waters.

Instead of adding magnesium supplements with a poor digestive tolerance, to patients with metastatic cancer and often with a heavy treatment , the aim of this study is to evaluate whether a change in oral hydration in quantitative and qualitative terms can decrease the rate of hypomagnesemia in patients treated with anti-EGFR.

ELIGIBILITY:
Inclusion Criteria:

1. Patient having either:

   * a metastatic head and neck cancer or in locoregional relapse, proved histologically, authorizing an oral feeding or by gastrostomy or nasogastric tube,
   * a metastatic colorectal cancer, histologically proved, wild-type RAS
2. Patient who must be treated by anti-EGFR for this cancer
3. Age ≥ 18 years
4. Performance Status = 0, 1 or 2
5. Patient affiliated to a social security scheme
6. Patient who have given written consent prior to any specific study-related procedure

Exclusion Criteria:

1. Cerebral metastasis
2. Previous anti-EGFR treatment
3. Patient requiring exclusive parenteral nutrition and hydration
4. Concomitant treatment by radiotherapy
5. Presence of another invasive cancer, other than head and neck or digestive, except basal cell carcinoma or intracervical neoplasia treated
6. Presence of hypomagnesemia at randomization
7. Ongoing oral or intravenous magnesium supplementation within 2 weeks before randomization
8. Patient with grade III or IV diarrhea within 2 weeks before randomization
9. Patient who have had a jejunostomy or ileostomy
10. Patient with constitutional tubulopathy
11. Patient with chronic renal insufficiency (MDRD Clarity <60 mL / min)
12. Pregnancy or breast-feeding
13. Persons deprived of their liberty or under guardianship
14. Dementia, mental impairment or psychiatric pathology that may compromise the patient's informed consent and / or adherence to the protocol and follow-up of the trial
15. Patient who can not follow protocol for psychological, social, family or geographical reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2023-01-04 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with hypomagnesemia | 3 months
  Determination of the blood magnesium level at each cycle

SECONDARY OUTCOMES:
Median rate of magnesium and hypomagnesemia grade III / IV | 6 months
  Determination of the blood magnesium level at each cycle
Proportion of patients with a 20% decrease in magnesemia | 6 months
  Determination of the blood magnesium level at each cycle
Incidence of hypomagnesemia after 2 cycles of anti-EGFR treatment | 6 months
  Determination of the blood magnesium level at each cycle
The fraction of urinary excretion over 24 hours of magnesium | 6 months
  Determination of urinary magnesium at the inclusion then at each even cycle of chemotherapy
Rate of patient requiring magnesium supplementation | 6 months
  Number of patient requiring magnesium supplementation (oral or IV)
Rate of hypomagnesemia at 5 months of treatment | 5 months
  Determination of the blood magnesium level at each cycle
Enteral intakes in magnesium | 6 months
  Completion of a feeding questionnaire at baseline and then at each even cycle. Completion of a patient notebook allowing daily monitoring of the quantity and type of water consumed Collection of concomitant treatment by magnesium
Quality of life | 6 months
  Completion of a quality of life questionnaire (QLQ-C30) at baseline and then at each even cycle
Compliance | 6 months
  Completion of a patient notebook allowing daily monitoring of the quantity and type of water consumed
Rate of diarrhea and cramps | 6 months
  Collection of adverse events classified according to NCI CTCAE V4.02
Hypocalcaemia and hypokalemia rates | 6 months
  Determination of blood calcium and potassium levels at the time of inclusion and then at each cycle of chemotherapy
Time until hypomagnesemia occurrence, regardless of grade, and time until grade III / IV hypomagnesemia | 6 months
  Time between treatment initiation and occurrence of hypomagnesemia
Progression-free survival | 2 years
  Time between treatment initiation and cancer progression
Overall survival | 2 years
  Time between treatment initiation and the patient's death within 2 years after treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Hugues BOURGEOIS, MD, Principal Investigator — Centre Jean Bernard - Le Mans
Locations (12):
- France (12):
  - GHBS Lorient, Lorient, Brittany Region
  - CARIO-HPCA Plérin, Plérin, Brittany Region
  - Centre Maurice TUBIANA, Caen, Normandy
  - CORT 37, Chambray-lès-Tours
  - Centre Hospitalier Départemental, La Roche-sur-Yon
  - Centre Hospitalier, Le Mans
  - Centre Jean Bernard, Le Mans
  - Polyclinique de Gentilly, Nancy
  - Centre Hospitalier, Niort
  - Centre Hospitalier Centre Bretagne, Pontivy
  - CHRU Tours, Tours
  - Centre d'Oncolgie Saint Yves, Vannes

IPD SHARING:
Plan to Share IPD: No